CLINICAL TRIAL: NCT06672679
Title: Juntos Latine Dating Violence Prevention Intervention Pilot
Brief Title: Juntos: A Pilot Test of a Dating Violence Intervention for Latine Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Maya Ragavan, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY24020165; K23HD104925 (NIH)
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-02

CONDITIONS: Intimate Partner Violence (IPV); Cultural Diversity; Prevention; Parent
Keywords: dating violence prevention; culturally affirming prevention; caregiver-adolescent intervention; Hispanic and Latino

STUDY DESIGN:
Intervention Model Description: We are using 3:1 recruitment (for every 3 intervention dyads, 1 control dyad) to ensure optimal investment in intervention group for this pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Juntos intervention (Experimental): In the Juntos intervention, 24 caregiver-adolescent dyads will receive a 6 week family-based dating violence prevention intervention called Juntos. Juntos includes 6 in-person sessions and 5 at home activities and was developed by Latino caregiver-adolescent dyads. Topics include cultural values and practices, talking about dating and dating violence, rule-setting, understanding signs of healthy and unhealthy relationships, and resources for support.
  Interventions: Behavioral: Juntos
- Control group (Active Comparator): The control arm will resource a resource guide and can be placed on a wait list to receive the intervention after the intervention is complete
  Interventions: Behavioral: Resource guide

INTERVENTIONS:
Behavioral: Juntos — 6 week family-based intervention
  Arms: Juntos intervention
Behavioral: Resource guide — Active control arm will receive a resource guide
  Arms: Control group

SUMMARY:
In this trial, we will be pilot-testing a family-based dating violence prevention program for Latine caregivers and adolescents. Participants will be randomized 1:1 to receive a community-based 6 week intervention or to a wait-list control where they will receive a resource guide.

ELIGIBILITY:
Inclusion Criteria:

Adolescents

1. Between the ages of 12-16
2. Identify as Hispanic or Latino/a/x/e
3. Speaks Spanish or English
4. Lives within 50 miles of Pittsburgh, Pennsylvania
5. Has a participating parent or caregiver* in the study

Adults

1. Over the age of 18
2. Identifies as Hispanic or Latino/a/x/e
3. Speaks Spanish
4. Lives within 50 miles of Pittsburgh, Pennsylvania
5. Is a caregiver of a participating adolescent in the study
6. Was born outside of the United States

Exclusion Criteria:

* Does not meet inclusion criteria
* Unable to consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Acceptability | weekly for 6 weeks, after each intervention session
  Acceptability Intervention Measure (scored on a Likert scale, 1 to 5 with 1 being completely disagree and 5 being completely agree). 4 items will be averaged for a summary score with higher numbers meaning higher acceptability.
Feasibility | baseline (pre-intervention), 1 week post-intervention follow up, 3 month post-intervention follow up surveys
  %participants who are enrolled, %consented, % randomized, % completed baseline, follow up and 3 month follow up surveys

SECONDARY OUTCOMES:
Self-efficacy in preventing dating violence | baseline (pre-intervention), 1 week post-intervention follow up, 3 month post-intervention follow up surveys
  11 item measure scored on a Likert scale to assess self-efficacy in preventing dating violence. Score for 7 items is on a 4 point Likert scale with 1: not at all confident and 4: very confident and the score for the other 3 items is 1 to 5 with 1: strongly disagree and 5: strongly agree. We will create a summary score which is the average of these 7 items, with higher numbers meaning higher self-efficacy around preventing dating violence.
Motivation to preventing dating violence | baseline (pre-intervention), 1-week post intervention follow up, 3 month post-intervention follow up surveys
  4 item measure scored on Likert scale focused on motivation caregivers and adolescents have around preventing dating violence. 0=not at all important and 10=very important. We will great a summary score which is an average of the 4 items, with a higher score indicating higher motivation around preventing dating violence.
Attitudes around dating violence | baseline (pre-intervention), 1-week post intervention follow up, 3 month post-intervention follow up surveys
  12 item measure assessing participants' attituding around dating violence scored on a Likert scale. 1: Not abusive: 2: a little abusive; 3: somewhat abusive; 4: very abusive; 5: extremely abusive. We will create a summary score which is an average of the 12 items, which higher scores indicating believing that the behaviors are more abusive
Caregiver-adolescent communication around dating violence | baseline (pre-intervention), 1-week post intervention follow up, 3 month post-intervention follow up surveys
  5 item measure scored on Likert scale assessing communication around dating violence. 0: never; 1: once; and 2: more than once. We will create a summary scare which is an average of the 5 items with higher numbers indicating more conversations.
Parental monitoring | baseline (pre-intervention), 1-week post intervention follow up, 3 month post-intervention follow up surveys
  Scale around dating and dating violence specific parental monitoring. This scale includes 6 items around time and resources scores on a 5 point Likert scale with 1: strongly disagree to 5: strongly agree; 2 items around parental knowledge of child's dating partner which is scored on a 5 point Likert scale with 1: strongly disagree and 5: strongly agree; 3 items around dating rule setting which is score on a 5 point Likert scale from 1: strongly disagree to 5: strongly agree and 4 items around child disclosure of dating violence scored on a 5 point Likert scale from 1:strongly disagree to 5; strongly agree. We will great a summary scale which is the average of the measures, with higher numbers indicating more parental monitoring.
Adolescent relationship abuse victimization (whether someone has experienced violence) | baseline (pre-intervention), 1-week post intervention follow up, 3 month post-intervention follow up surveys
  25 item measure to assess experiences of physical, emotional, sexual, economic, and digital dating violence (0=never experienced; 1=experienced but not in the last year; and 2=experienced in the last year)
Adolescent relationship abuse perpetration (whether someone has used violence) | baseline (pre-intervention), 1-week post intervention follow up, 3 month post-intervention follow up surveys
  25 item measure to assess experiences of physical, emotional, sexual, economic, and digital dating violence perpetration (0=never experienced; 1=experienced but not in the last year; and 2=experienced in the last year)

OTHER OUTCOMES:
Ethnic Identity | baseline (pre-intervention), 1-week post intervention follow up, 3 month post-intervention follow up surveys
  Multiethnic Identity Measure; 12 item scale on a 4 point Likert scale from 1: strongly disagree to 4: strongly agree. Summary score of the average of 12 items with higher scores indicating more ethnic identity.
Acculturation conflict measure | baseline (pre-intervention), 1-week post intervention follow up, 3 month post-intervention follow up surveys
  7 item acculturation conflict measure (investigator developed) scored on a 4 point Likert Scale from 1: strongly disagree to 4: strongly agree. A summary score of the average of the 7 items will be computed, with higher scores indicating more parent-adolescent acculturation conflict.
Discrimination Scale | baseline (pre-intervention), 1-week post intervention follow up, 3 month post-intervention follow up surveys
  9 item Everyday Discrimination Scale scored on a 6 point Likert scale with 1: never to 6: every day. A summary score (average of the 9 items) will be created with higher scores indicating more experiences of discrimination.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Primary Care Center, Pittsburgh, Pennsylvania
  - Casa San Jose, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Due to the sensitivity of the survey data, we will not share individual patient data